CLINICAL TRIAL: NCT04227210
Title: A Phase 1 Study to Evaluate the Safety and Immunogenicity of an Intranasal Live Attenuated Respiratory Syncytial Virus (RSV) Vaccine in Healthy Adults
Brief Title: Safety and Immune Response to an Investigational Vaccine Against Respiratory Syncytial Virus in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meissa Vaccines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MV-003
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: vaccine; live attenuated; safety; immunogenicity; viral shedding; phase 1 clinical trial
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Each enrolled subject will be allocated to 1 of 2 study groups. Group 1 will receive one dosage of the investigational RSV vaccine, and Group 2 will receive a different dosage of the same vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSV Vaccine: Dosage Group #1 (Experimental): Participants in this group will receive a single dose of the RSV vaccine at dosage #1
  Interventions: Biological: RSV vaccine MV-012-968 (dosage #1)
- RSV Vaccine: Dosage Group #2 (Experimental): Participants in this group will receive a single dose of the RSV vaccine at dosage #2
  Interventions: Biological: RSV vaccine MV-012-968 (dosage #2)

INTERVENTIONS:
Biological: RSV vaccine MV-012-968 (dosage #1) — Single dose administered intranasally on Day 1
  Arms: RSV Vaccine: Dosage Group #1
Biological: RSV vaccine MV-012-968 (dosage #2) — Single dose administered intranasally on Day 1
  Arms: RSV Vaccine: Dosage Group #2

SUMMARY:
This study evaluates an investigational vaccine designed to protect humans against infection with respiratory syncytial virus (RSV). The investigational vaccine (MV-012-968) is administered as drops in the nose. This study specifically analyzes the safety of, and the immune response to, the vaccine when administered to healthy non-pregnant adults between the ages of 18 and 40 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult 18-40 years of age
* In good health based on review of the medical record, history, and physical examination, without evidence of chronic disease
* RSV 'sero-low' from a pre-vaccination serum sample
* Signed informed consent form

Exclusion Criteria:

* Occupational or household exposure to children < 5 years of age, or to immunocompromised individuals
* Prior receipt of an investigational RSV vaccine
* Women who are pregnant, lactating, or unwilling to take effective measures to prevent pregnancy for at least 3 months after vaccination
* Any other reason the Investigator considers exclusionary

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events (AEs) | Immediate post-vaccination period
  Frequency of solicited AEs will be measured, categorized by severity. Solicited AEs are predefined AEs that can occur after vaccine administration.
Unsolicited AEs | Immediate post-vaccination period
  Frequency of unsolicited AEs will be measured, categorized by severity. Unsolicited AEs are any untoward medical occurrences in a participant administered the investigational vaccine, regardless of causal relationship to the investigational vaccine. Unsolicited AEs can include unfavorable and unintended signs (including abnormal laboratory findings), symptoms, or diseases temporally associated with the use of the investigational vaccine.
Serious adverse events (SAEs) | Vaccination through study completion, an average of 6 months
  Frequency of SAEs will be measured, categorized by vaccine-relatedness. SAEs are AEs, whether considered causally related to the investigational vaccine or not, that threaten life or result in any of the following: death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or congenital anomaly/birth defect.
Medically attended adverse events (MAEs) | Vaccination through study completion, an average of 6 months
  Frequency of MAEs will be measured, categorized by vaccine-relatedness. MAEs are AEs, whether considered causally related to the investigational vaccine or not, with unscheduled medically attended visits, such as urgent care visits, acute primary care visits, emergency department visits, or other previously unplanned visits to a medical provider. Scheduled medical visits such as routine physicals, wellness checks, 'check-ups', and vaccinations, are not considered MAEs.

SECONDARY OUTCOMES:
Change in serum RSV-specific neutralizing antibody (nAb) titers | Baseline through study completion, an average of 6 months
  Post-vaccination change in serum RSV-specific nAb titers will be measured per participant.
Change in serum RSV F-specific binding antibody titers | Baseline through study completion, an average of 6 months
  Post-vaccination change in serum RSV F-specific binding antibody titers will be measured per participant.
Change in mucosal RSV F-specific binding antibody titers | Baseline through study completion, an average of 6 months
  Post-vaccination change in mucosal RSV F-specific binding antibody titers will be measured per participant.
Potential vaccine virus shedding | Baseline through 2 months
  The presence and, if detected, quantity and duration of any shed vaccine virus will be measured per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Medzihradsky, MD MPH MS, Study Director — Meissa Vaccines, Inc.
Locations (1):
- Johnson County Clin-Trials, Lenexa, Kansas, United States

REFERENCES:
- [Background] Stobart CC, Rostad CA, Ke Z, Dillard RS, Hampton CM, Strauss JD, Yi H, Hotard AL, Meng J, Pickles RJ, Sakamoto K, Lee S, Currier MG, Moin SM, Graham BS, Boukhvalova MS, Gilbert BE, Blanco JC, Piedra PA, Wright ER, Moore ML. A live RSV vaccine with engineered thermostability is immunogenic in cotton rats despite high attenuation. Nat Commun. 2016 Dec 21;7:13916. doi: 10.1038/ncomms13916. PMID 28000669